CLINICAL TRIAL: NCT00934596
Title: CO2 Insufflation vs Lund De-airing Technique For Open Left Heart Surgery - Safety and Efficacy
Brief Title: CO2 Versus Lund De-airing Technique in Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Bansi Lal Koul, Chief Surgeon and Associate Professor, Lund University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Lund de-airing technique
Record Dates: First submitted 2009-07-07; First posted 2009-07-08 (Estimated); Results first posted 2013-12-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-10

CONDITIONS: Aortic Valve Disorder
Keywords: Cardiac de-airing; CO2 insufflation; Air emboli; Trans cranial doppler; Intraoperative echocardiography
MeSH Terms: conditions — Aortic Valve Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lund de-airing (Experimental): Lund de-airing technique
  Interventions: Procedure: Lund de-airing technique
- Carbon-dioxide insufflation (Active Comparator): carbon-dioxide insufflation will be provided to the open mediastinal wound in a standardized manner
  Interventions: Drug: carbon-dioxide insufflation

INTERVENTIONS:
Procedure: Lund de-airing technique — In these patients the pleura will be opened on both sides and the ventilator will be disconnected before aorta is cross-clamped and cardioplegia administered. At the conclusion of the surgical procedure, the LV preload will first now be successively increased. When no air is seen on TEE monitoring in the left heart (LA, LV & Aorta), half the calculated minute ventilation with 100% oxygen and a PEEP of 5 cm H2O will be started. Deairing will be continued and when the TEE shows no or minimal air in left heart, full ventilation with unchanged PEEP will be restored. The patient will be weaned successively from the CPB. When TEE will show no air in the left heart, the de-airing will be considered complete.
  Other Names: cardiac de-airing; cardiac venting
  Arms: Lund de-airing
Drug: carbon-dioxide insufflation — In these patients (n=10) the pleurae will not be opened. During aortic cross-clamp period the ventilator will be adjusted to provide dead space ventilation only i.e. 5cm PEEP, ventilator frequency 5/min and the minute ventilation = 1,5 liter. Fio2 = 50%. The operating field will be insufflated with Co2 at a flow rate of 10 L / minute starting 2 minutes before cardiac cannulation and continued until 10 minutes after termination of the CPB.At the end of the cardioplegic arrest, the de-airing procedure is similar to that in the Lund de-airing group.
  Other Names: Cardiac de-airing; Cardiac venting
  Arms: Carbon-dioxide insufflation

SUMMARY:
To evaluate which of the two de-airing methods (CO2 insufflation vs. Lund de-airing technique) can shorten the left heart de-airing time and prevent or minimize cerebral air emboli during open surgery involving exposure of the left heart to the ambient air.

To evaluate the cost effectiveness and possible side effects of CO2 de-airing technique compared to Lund de-airing technique.

DETAILED DESCRIPTION:
Study design:

Prospective, randomized and controlled study involving 20 patients, 10 in each group. The de-airing time and the efficiency of the techniques will be assessed by trans-esophageal echocardiography (TEE) and trans-cranial echo-doppler monitoring (TCD). The cardiologists analyzing the TEE recordings will be blinded to the de-airing technique used (the recorded videos will be analyzed at the end of the study). The TCD monitoring will be done by on-line automatic recording of the micro embolic signals (MES) from the right and or left middle cerebral arteries and performed by single surgeon. The CO2 insufflation of the operating field will be performed according to manufacturer's guide lines. During entire study course one type of extracorporeal perfusion system will be used.The study will be registered in the international database. A prior approval will be sought from the hospital ethical committee for the study.

Patient selection:

Patients planned for aortic valve/root replacement or repair will be selected for the study

Exclusion criteria:

Patients with known: a) chronic obstructive pulmonary disease, b) emphysema, c) previous thoracic or cardiac surgery, d) history of CVA or stroke and e) evidence of intraoperative pleural adhesions will be excluded from the study. Patients requiring internal mammary artery coronary bypass will also be excluded.

Patient consent:

A written consent previously approved by the hospital ethical committee will be obtained from all patients before they are enrolled in the study (enclosure 3).

De-airing procedure:

Enrolled patients will be assigned randomly to one of the two following groups:

Control group ( newly developed de-airing technique in Lund ) :

In these patients (n=10) the pleura will be opened on both sides and the ventilator will be disconnected before aorta is cross-clamped and cardioplegia administered. At the end of the cardioplegic arrest, the aortic root and the LV will be actively vented and aortic cross clamp released. The time will be noted down (T1). The heart will be defibrillated to sinus or pacemaker induced rhythm. The heart will be kept empty by the LV vent and ejection avoided as monitored by continual intraoperative TEE and systemic arterial pressure tracing. At 35 Celsius body temperature, as measured from the thermistor in the urinary bladder, and with apparently good cardiac contraction the de-airing will begin. Inotropic drugs or systemic arterial vasodilators will be used as and when necessary to achieve good cardiac contraction. The time will be noted down (T2) (T2 - T1 = Pre ejection de-airing time). The LV preload will first now be successively increased by reducing the venous return from the heart-lung machine to raise CVP between 5-10 cm water. LV vent will be continuously regulated depending upon the amount of residual air showing in the left heart. When no air is seen on TEE monitoring in the left heart (LA, LV & Aorta), half the calculated minute ventilation with 100% oxygen and a PEEP of 5 cm H2O will be started. De-airing will be continued and when the TEE shows no or minimal air in left heart, full ventilation with unchanged PEEP will be restored. The patient will be weaned successively from the CPB thereby ensuring that entire cardiac output is diverted through the native fully ventilated lungs. When TEE will show no air in the left heart, the de-airing will be considered complete and the time noted again (T3) (T3 - T2 = Post ejection de-airing time).

All cardiac cannulae including the LV vent will be left in situ but clamped, patient weaned completely from the cardiopulmonary bypass and monitored for residual air by TEE & TCD for 10 minutes continually. The LV vent will be re-opened whenever the residual air in the left heart exceeds grade II. The frequency of theses measures will be noted in the protocol. If the patient has by now achieved 36 Celsius core temperature, the heart will be decannulated and CPB removed. Otherwise CPB will be restarted and patient warmed to 36 Celsius before final weaning and decannulation.

Study group ( CO2 insufflation ):

In these patients (n=10) the pleurae will not be opened. During aortic cross-clamp period the ventilator will be adjusted to provide dead space ventilation only i.e. 5cm PEEP, ventilator frequency 5/min and the minute ventilation = 1,5 liter. Fio2 = 50%. The operating field will be insufflated with CO2 at a flow rate of 10 L / minute starting 2 minutes before cardiac cannulation and continued until 10 minutes after termination of the CPB.

At the end of the cardioplegic arrest, the aortic root and the LV will be actively vented and the time noted down (T1). The LV preload will be successively increased by reducing the venous return from the heart-lung machine to raise CVP between 5-10 cm water. LV venting will be continued and when no air bubbles are seen in the left heart (LA, LV & Aorta) under TEE monitoring, the calculated minute ventilation with 100% oxygen and PEEP of 5 cm H2O will be restored. De-airing will be continued and when no or minimal air is seen in the left heart the time will be noted down (T2) (T2 - T1 = Pre ejection de-airing time). Aortic cross-clamp will be released now and heart defibrillated to sinus or pacemaker induced rhythm and de-airing continued. At 35 Celsius body temperature, as measured from the thermistor in the urinary bladder, and with apparently good cardiac contraction the patient will be weaned successively from the CPB ensuring thereby that the entire cardiac output is diverted through the native fully ventilated lungs. Inotropic drugs or systemic arterial vasodilators will be used as and when necessary to achieve good cardiac contraction. When TEE will show no air in the left heart, the de-airing will be considered complete and the time noted again (T3) (T3 - T2 = Post ejection de-airing time). The patient will be weaned completely from the cardiopulmonary bypass and all cardiac cannulae including the LV vent will be left in situ but clamped. The patient will be monitored now for residual air by TEE & TCD for 10 minutes continually. The LV vent will be re-opened whenever the residual air showing on TEE in the left heart exceeds grade II. The frequency of theses measures will be noted in the protocol. The C02 insufflations will continue until the 10- minute post CPB monitoring interval is completed. If patient by now has achieved 36 Celsius core temperature, the heart will be decannulated and CPB removed. Otherwise CPB will be restarted and patient warmed to 36 Celsius before final weaning and decannulation.

Trans-esophageal echocardiographic study (TEE):

After completion of the cardioplegic arrest and for 10 minutes after termination of the CPB, all the patients will be monitored by TEE for air in the left heart. The residual air showing on TEE after the termination of CPB will be quantified in 4 grades depending upon presence of air in LA, LV and aortic root during one cardiac cycle (grade 0 = no or occasional air in LA, grade 1 = air showing in LA only, grade 2 = air showing simultaneously in LA and LV, grade 3 = air showing simultaneously in LA, LV and the aortic root). The 10-minute post CPB TEE recording will be saved on a video-tape.

Trans-cranial echo-doppler study (TCD):

After release of the aortic cross clamp and for 10 minutes after the patient has been weaned off from the CPB, the patient will be continuously monitored for micro embolic signals by on-line automatic TCD placed on middle cerebral arteries.

Blood gases will be monitored in all patients as following:

Blood gas analysis from arterial & venous blood of the patient every 15 minutes in the operating room in both groups until 15 minutes post CPB) - following attached tables (Anesthesia, Perfusion and TCD & Invous monitoring)

Measurement of end-tidal PCO2 and volume of expired CO2 every 15 minutes after the patient is intubated and till the time patient leaves the operating room in both groups. (No measurements possible in the control group during cardioplegic arrest)

Blood gas analysis from arterial & venous blood lines of the oxygenator and from the LV vent line every 15 minutes while the patient is on CPB in both groups.

Continuous on-line monitoring of CO2 content and PCO2 in the blood at the inflow and outflow ports of the oxygenator in both groups using CDI & new machine. Variations in gas flow and the FiO2 needed to adjust PaCO2 to within a fixed desirable range will be recorded and extra blood gas sample will be taken whenever any such adjustment is made.

Alfa stat will be employed for blood gas analysis. A core temperature at 30 C will be used for all patients unless positively indicted.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for aortic valve/root replacement or repair will be selected for the study

Exclusion Criteria:

Patients with known

* chronic obstructive pulmonary disease,
* emphysema,
* previous thoracic or cardiac surgery,
* history of CVA or stroke and
* evidence of intraoperative pleural adhesions will be excluded from the study.
* Patients requiring internal mammary artery coronary bypass will also be excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bansi L Koul, MD, PhD, Principal Investigator — Cardiothoracic Surgery, Heart & Lung Division, University Hospital Lund, Sweden

REFERENCES:
- [Derived] Landenhed M, Al-Rashidi F, Blomquist S, Hoglund P, Pierre L, Koul B. Systemic effects of carbon dioxide insufflation technique for de-airing in left-sided cardiac surgery. J Thorac Cardiovasc Surg. 2014 Jan;147(1):295-300. doi: 10.1016/j.jtcvs.2012.11.010. Epub 2012 Dec 13. PMID 23246060
- [Derived] Al-Rashidi F, Landenhed M, Blomquist S, Hoglund P, Karlsson PA, Pierre L, Koul B. Comparison of the effectiveness and safety of a new de-airing technique with a standardized carbon dioxide insufflation technique in open left heart surgery: a randomized clinical trial. J Thorac Cardiovasc Surg. 2011 May;141(5):1128-33. doi: 10.1016/j.jtcvs.2010.07.013. Epub 2010 Sep 3. PMID 20817209

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients requiring elective aortic valve or aortic root surgery on the waiting list of the clinic were recruited in the study during year 2009.
Pre-assignment Details: All 20 consecutive patients recruited in the study fullfilled the inclusion criteria. No patient was excluded.
Groups:
- Lund De-airing Technique: Before cardiopulmonary bypass (CPB) was established, both pleural cavities were exposed to atmospheric air through small openings in the mediastinal pleurae. After CPB was established the patient was disconnected from the ventilator, allowing both lungs to collapse. After completion of the surgical procedure the aortic crossclamp was released and the heart was then defibrillated. After a good cardiac contraction and normal central hemodynamics, the LV preload was gradually and successively. When no air emboli were observed in the left side of the heart by Trans-esophageal Echocardiography (TEE), the patient was reconnected to the ventilator and the lungs were ventilated with half of the estimated minute volume using 100% oxygen and 5 cm H2O positive end-expiratory pressure. The de-airing was continued, and when no air emboli were observed in the left side of the heart, the lungs were ventilated to full capacity and the heart was allowed to eject by reducing the LV vent.
- Carbon-dioxide Insufflation Technique: The pleural cavities were left intact in the carbon-dioxide(CO2) group. During cardiopulmonary bypass (CPB), the patient was administered dead space ventilation. Before the cannulation for CPB, the CO2 was insufflated in the mediastinum at a flow rate of 10 L/min and continued until 10 minutes post-CPB. After completed surgery, the heart and lungs were passively filled with blood from the CPB circuit and the left side was de-aired continuously through the LV apical vent. Full ventilation was then resumed. The heart was defibrillated and the LV preload was gradually and successively increased by reducing the venous return to the CPB circuit. The de-airing continued through the vent in the LV apex under TEE monitoring. When no gas emboli were observed in the left side of the heart, the LV vent was reduced and the heart was allowed to ject. De-airing was continued, and when no further gas emboli were observed in the left side of the heart, the patient was weaned from CPB.
Period: Overall Study
Arm/Group | Lund De-airing Technique | Carbon-dioxide Insufflation Technique
Started | 10 (Twenty patients were prospectively randomly assigned to the two arms) | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Lund De-airing Technique: Before cardiopulmonary bypass (CPB) was established, both pleural cavities were exposed to atmospheric air through small openings in the mediastinal pleurae. Hereafter the patient was disconnected from the ventilator, allowing both lungs to collapse. After completion of the surgical procedure the aortic crossclamp was released and the heart defibrillated. After a good cardiac contraction and normal central hemodynamics were established, the LV preload was gradually and successively increased. When no air emboli were observed in the left side of the heart by transesophageal echocardiography (TEE), the patient was reconnected to the ventilator and the lungs were ventilated with half of the estimated minute volume using 100% oxygen and 5 cm H2O positive end-expiratory pressure. The deairing was continued, and when no air emboli were observed in the left side of the heart, the lungs were ventilated to full capacity and the heart was allowed to eject by reducing the LV vent.
- Carbon-dioxide Insufflation Technique: The pleural cavities were left intact in the CO2 (carbon-dioxide) group. During cardiopulmonary bypass (CPB), the patient was administered dead space ventilation. Before cannulation, CO2 was insufflated in the mediastinum at a flow rate of 10 litres/minute and continued until 10 minutes post-CPB. After completed surgery, the heart and lungs were passively re-filled with blood and the left side was de-aired continuously through the LV apical vent. Full ventilation was then resumed. The heart was defibrillated and the LV preload was gradually and successively increased by reducing the venous return to the CPB circuit. The de-airing continued through the vent in the LV apex under transesophageal echocardiographic (TEE) monitoring. When no gas emboli were observed in the left side of the heart, the LV vent was reduced and the heart was allowed to eject. De-airing was continued, and when no further gas emboli were observed in the left side of the heart, the patient was weaned from CPB.
- Total: Total of all reporting groups
Arm/Group | Lund De-airing Technique | Carbon-dioxide Insufflation Technique | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 9 | 7 | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 68 (11) | 68 (13) | 68 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  Sweden | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Air Microemboli Registered Over the Middle Cerebral Arteries by On-line Trans-cranial Echo-Doppler (TCD).
Description: The number of air microemboli (also referred to as gaseous microembolic signals) was concomitantly counted in the right and left medial cerebral artery. The number of signals from the right and the left medial cerebral artery were summed, and presented as the total sum of the gaseous micromebolic signals from the right and left side. Counting of gaseous microembolic signals was done during three time intervals: Before cardiac ejection, after cardiac ejection and during 10 minutes after cardiopulmonary bypass.
Time Frame: Before cardiac ejection
Measure: Mean (Standard Deviation); unit: Air Microemboli
Groups:
- Lund De-airing Technique: Before cardiopulmonary bypass(CPB) was started, both pleural cavities were exposed to atmospheric air through small openings in the mediastinal pleurae. After CPB was established the patient was disconnected from the ventilator, allowing both lungs to collapse. After completion of the surgical procedure the aortic crossclamp was released and the heart was then defibrillated. After a good cardiac contraction and normal central hemodynamics, the LV preload was gradually and successively. When no air emboli were observed in the left side of the heart, the patient was reconnected to the ventilator and the lungs were ventilated with half of the estimated minute volume using 100% oxygen and 5 cm H2O positive end-expiratory pressure. The de-airing was continued, and when no air emboli were observed in the left side of the heart, the lungs were ventilated to full capacity and the heart was allowed to eject by reducing the LV vent.
- Carbon-dioxide Insufflation Technique: The pleural cavities were left intact in the CO2 (carbon-dioxide) group. During cardiopulmonary bypass (CPB), the patient was administered dead space ventilation. Before CPB, the CO2 was insufflated in the mediastinum at a flow rate of 10 L/min and continued until 10 minutes post-CPB. After completion of the surgical procedure, the heart and lungs were passively filled with blood from the CPB circuit and the left side was de-aired continuously through the LV apical vent. Full ventilation was then resumed. The heart was defibrillated and the LV preload was gradually and successively increased by reducing the venous return to the CPB circuit. The de-airing continued through the vent in the LV apex under TEE monitoring. When no gas emboli were observed in the left side of the heart, the LV vent was reduced and the heart was allowed to ject. De-airing was continued, and when no further gas emboli were observed in the left side of the heart, the patient was weaned from C
Arm/Group | Lund De-airing Technique | Carbon-dioxide Insufflation Technique
Number analyzed (Participants) | 10 | 10
Air Microemboli | 41 (20) | 118 (70)
Statistical Analysis 1: Comparison: Lund De-airing Technique vs Carbon-dioxide Insufflation Technique; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney); Median Difference (Net) = 57

2. Secondary Outcome: Total Time Required for De-airing
Description: The total de-airing time as measured in minutes.
Time Frame: After removal of aortic cross-clamp to complete de-airing, an average of 11 minutes
Measure: Median (Inter-Quartile Range); unit: Minutes
Groups:
- Lund De-airing Technique: Before CPB was started, both pleural cavities were exposed to atmospheric air through small openings in the mediastinal pleurae. After CPB was established the patient was disconnected from the ventilator, allowing both lungs to collapse. After completion of the surgical procedure the aortic crossclamp was released and the heart was then defibrillated. After a good cardiac contraction and normal central hemodynamics, the LV preload was gradually and successively. When no air emboli were observed in the left side of the heart, the patient was reconnected to the ventilator and the lungs were ventilated with half of the estimated minute volume using 100% oxygen and 5 cm H2O positive end-expiratory pressure. The deairing was continued, and when no air emboli were observed in the left side of the heart, the lungs were ventilated to full capacity and the heart was allowed to eject by reducing the LV vent.
- Carbon-dioxide Insufflation Technique: The pleural cavities were left intact in the CO2 group. During CPB, the patient was administerd dead space ventilation. Before the cannulation for CPB, the CO2 was insufflated in the mediastinum at a flow rate of 10 L/min and continued until 10 minutes post-CPB. After completion of the surgical procedure, the heart and lungs were passively filled with blood from the CPB circuit and the left side was de-aired continuously through the LV apical vent. Full ventilation was then resumed. The heart was defibrillated and the LV preload was gradually and successively increased by reducing the venous return to the CPB circuit. The de-airing continued through the vent in the LV apex under TEE monitoring. When no gas emboli were observed in the left side of the heart, the LV vent was reduced and the heart was allowed to ject. De-airing was continued, and when no further gas emboli were observed in the left side of the heart, the patient was weaned from CPB.
Arm/Group | Lund De-airing Technique | Carbon-dioxide Insufflation Technique
Number analyzed (Participants) | 10 | 10
Minutes | 9 [8 to 10] | 15 [11 to 16]

3. Secondary Outcome: De-airing Time Before Cardiac Ejection
Description: Time in minutes starting at t1 (removal of aortic cross clamp) and ending at t2 (beginning of cardiac ejection).
Time Frame: Measured during intraoperative course
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- Lund De-airing: Before CPB was started, both pleural cavities were exposed to atmospheric air through small openings in the mediastinal pleurae. After CPB was established the patient was disconnected from the ventilator, allowing both lungs to collapse. After completion of the surgical procedure the aortic crossclamp was released and the heart was then defibrillated. After a good cardiac contraction and normal central hemodynamics, the LV preload was gradually and successively. When no air emboli were observed in the left side of the heart, the patient was reconnected to the ventilator and the lungs were ventilated with half of the estimated minute volume using 100% oxygen and 5 cm H2O positive end-expiratory pressure. The deairing was continued, and when no air emboli were observed in the left side of the heart, the lungs were ventilated to full capacity and the heart was allowed to eject by reducing the LV vent.
- Carbon-dioxide Insufflation: The pleural cavities were left intact in the CO2 group. During CPB, the patient was administerd dead space ventilation. Before the cannulation for CPB, the CO2 was insufflated in the mediastinum at a flow rate of 10 L/min and continued until 10 minutes post-CPB. After completion of the surgical procedure, the heart and lungs were passively filled with blood from the CPB circuit and the left side was de-aired continuously through the LV apical vent. Full ventilation was then resumed. The heart was defibrillated and the LV preload was gradually and successively increased by reducing the venous return to the CPB circuit. The de-airing continued through the vent in the LV apex under TEE monitoring. When no gas emboli were observed in the left side of the heart, the LV vent was reduced and the heart was allowed to ject. De-airing was continued, and when no further gas emboli were observed in the left side of the heart, the patient was weaned from CPB.
Arm/Group | Lund De-airing | Carbon-dioxide Insufflation
Number analyzed (Participants) | 10 | 10
minutes | 6 [4 to 7] | 7 [5 to 10]

4. Primary Outcome: Number of Air Microemboli Registered Over the Middle Cerebral Arteries by On-line Trans-cranial Echo-Doppler (TCD).
Description: as for outcome 1
Time Frame: After cardiac ejection
Measure: Mean (Standard Deviation); unit: Air Microemboli
Arm/Group | Lund De-airing Technique | Carbon-dioxide Insufflation Technique
Number analyzed (Participants) | 10 | 10
Air Microemboli | 28 (19) | 119 (84)
Statistical Analysis 1: Comparison: Lund De-airing Technique vs Carbon-dioxide Insufflation Technique; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Net) = 72

5. Secondary Outcome: De-airing Time After Cardiac Ejection
Description: The duration in minutes of the period after cardiac ejection to finished de-airing procedure.
Time Frame: During de-airing procedure
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Lund De-airing | Carbon-dioxide Insufflation
Number analyzed (Participants) | 10 | 10
minutes | 3 [2 to 3] | 5 [4 to 8]

6. Secondary Outcome: Oxygenator Gas Flow at 45 Minutes of CPB
Description: The amount of carbon dioxide gas flow through the oxygenator was measured and compared between groups.
Time Frame: Intraoperative
Measure: Median (Inter-Quartile Range); unit: L/minute
Arm/Group | Lund De-airing | Carbon-dioxide Insufflation
Number analyzed (Participants) | 10 | 10
L/minute | 0.65 [0.60 to 1.25] | 2.2 [1.63 to 3.10]

7. Post Hoc Outcome: Fraction of Morphologically Damaged Red Blood Cells as Assessed by Scanning Electron Microscopy Studies.
Description: Pieces of tubing from the cardiopulmonary circuit were prepared and photographed in a Scanning Electron Microscope. Visual inspection of each photograph by an investigator blinded to which group the photograph belonged to was performed. The proportion of damaged red blood cells over the total number of red blood cells were calculated.
Time Frame: Pieces of tubing collected after weaning from cardiopulmonary bypass
Population: Samples were collected from 5 participants in each Group (total of 10 participants). For each participant 4 pieces of tubing were collected (20 pieces in each Group, total 40 pieces). Samples were photographed. One photograph from each individual was randomly selected and studied by an investigator blinded to Group (total of 10 photographs).
Measure: Mean (95% Confidence Interval); unit: Fraction of Damaged Red Blood Cells
Arm/Group | Lund De-airing Technique | Carbon-dioxide Insufflation Technique
Number analyzed (Participants) | 5 | 5
Fraction of Damaged Red Blood Cells | 0.18 [0.11 to 0.30] | 0.97 [0.64 to 1.0]

8. Secondary Outcome: pH at 45 Min of CPB
Description: pH measured by arterial bloodgas at 45 minutes of CPB, comparison between groups
Time Frame: Intraoperative
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Lund De-airing | Carbon-dioxide Insufflation
Number analyzed (Participants) | 10 | 10
units on a scale | 7.30 [7.27 to 7.33] | 7.35 [7.32 to 7.38]

9. Primary Outcome: Number of Air Microemboli Registered Over the Middle Cerebral Arteries by On-line Trans-cranial Echo-Doppler (TCD).
Description: as for outcome 1
Time Frame: During 10 minutes after cardiopulmonary bypass
Measure: Mean (Standard Deviation); unit: Air Microemboli
Arm/Group | Lund De-airing Technique | Carbon-dioxide Insufflation Technique
Number analyzed (Participants) | 10 | 10
Air Microemboli | 5 (4) | 46 (53)
Statistical Analysis 1: Comparison: Lund De-airing Technique vs Carbon-dioxide Insufflation Technique; As data for these small groups were non-parametric the median and quartiles were used for comparison of groups by the Wilcoxon Rank Sum test; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney); Median Difference (Net) = 17

10. Primary Outcome: Number of Participants With <=Grade I Gas Emboli as Assessed by Trans-esophageal Echocardiography TEE).
Description: Grade 0, no residual gas emboli; grade I, gas emboli observed in 1 of the 3 anatomic areas - left atrium, left ventricle or aortic root during 1 cardiac cycle; grade II, gas emboli observed simultaneously in 2 of the 3 anatomic areas during 1 cardiac cycle; grade III, gas emboli observed simultaneously in all 3 anatomic areas during 1 cardiac cycle.
Time Frame: 0-3 minutes after end of cardiopulmonary bypass
Population: The number was determined before hand as per protocoll.
Measure: Number; unit: participants
Arm/Group | Lund De-airing Technique | Carbon-dioxide Insufflation Technique
Number analyzed (Participants) | 10 | 10
participants | 10 (4) [25 to 75] | 4 (53) [25 to 75]

11. Primary Outcome: Number of Participants With <=Grade I Gas Emboli as Assessed by Trans-esophageal Echocardiography TEE).
Description: as for outcome 10
Time Frame: 3-6 minutes after end of cardiopulmonary bypass
Population: The number was determined before hand as per protocoll.
Measure: Number; unit: participants
Arm/Group | Lund De-airing Technique | Carbon-dioxide Insufflation Technique
Number analyzed (Participants) | 10 | 10
participants | 9 | 7

12. Primary Outcome: Number of Participants With <=Grade I Gas Emboli as Assessed by Trans-esophageal Echocardiography TEE).
Description: as for outcome 10
Time Frame: 6-10 minutes after end of cardiopulmonary bypass
Population: The number was determined before hand as per protocoll.
Measure: Number; unit: participants
Arm/Group | Lund De-airing Technique | Carbon-dioxide Insufflation Technique
Number analyzed (Participants) | 10 | 10
participants | 9 | 7

ADVERSE EVENTS:
Time Frame: Data was collected during the postoperative course when patient was still in ward (median time 7 Days).
Description: Method of detecting adverse events was screening of patients charts for reports of neurological dysfunction.
Arm/Group | Lund De-airing | Carbon-dioxide Insufflation
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lund De-airing (N=10) | Carbon-dioxide Insufflation (N=10)
Postoperative neurological dysfunction (Nervous system disorders) | 1 (1) | 1 (1) — Any sign of postoperative confusion, agitation or disorientation OR focal neurological deficit with or without cerebral computer tomography performed.

LIMITATIONS AND CAVEATS:
This study included a total of 20 patients randomized to one of two groups with ten patients in each arms. The small number of study objects might be a potential limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No